CLINICAL TRIAL: NCT02604927
Title: Beta-alanine Supplementation and Its Effects on Performance, Muscle Carnosine Content and Safety in Athletes With Spinal-cord Injury
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Bruno Gualano, Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: B-Alanine Paraplegic Athletes
Record Dates: First submitted 2015-09-22; First posted 2015-11-16 (Estimated); Last update posted 2015-11-16 (Estimated); Status verified 2015-11

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries | interventions — beta-Alanine; Glucose

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): 800 mg of dextrose, four times per day, during 28 days.
  Interventions: Dietary Supplement: Dextrose
- Beta-alanine (Experimental): 800 mg of beta-alanine, four times per day, during 28 days.
  Interventions: Dietary Supplement: Beta-alanine

INTERVENTIONS:
Dietary Supplement: Beta-alanine
  Arms: Beta-alanine
Dietary Supplement: Dextrose
  Arms: Placebo

SUMMARY:
Paralympians competing in wheelchair sports may experience a very high glycolytic demand (and therefore acidotic environment) in their upper-body muscles, particularly in high-intensity disciplines. Previous studies from our group have shown that upper-body exercise is very sensitive to the ergogenic effects of β-alanine supplementation and to other nutritional supplements capable of increasing buffering capacity. In line with this, have shown that upper-body muscle groups benefit more from artificially induced alkalosis than lower-body muscle groups. Although β-alanine appears to be an interesting and potential ergogenic supplement for paralympians, no study to date has assessed its potential in wheelchair athletes.In this study, we will evaluate the effects of β-alanine supplementation on upper-body performance in wheelchair athletes.

ELIGIBILITY:
Inclusion Criteria:

* Paralympian training for any exercise modality for at least one year;
* A weekly training volume of 6 hours or more;
* Have a spinal cord injury accompanied by loss of motor function in the lower limbs for at least one year;
* Available for carrying out the experimental procedures.

Exclusion Criteria:

* Use of creatine or beta-alanine for at least 3 and 6 months before the trial;
* Cardiovascular or respiratory disease;
* Clinical condition that result in malabsorption of nutrients;
* Any other medical condition that prevents the realization of experimental procedures.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-02; Primary Completion 2016-11 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Exercise performance (Time to exhaustion test) | 28 days
  Time to exhaustion test performed on arm crank ergometer
Muscle carnosine content before and after supplementation | 28 days
  Assessed by muscle biopsy samples before performance tests

SECONDARY OUTCOMES:
Muscle carnosine content in trained (deltoid) vs. untrained (vastus lateralis) muscles | 28 days
  Deltoids microbiopsy and vastus lateralis biopsy
Blood pH. | 5 minutes after performance tests
  1 mL venous blood sample
Safety of beta-alanine supplementation measured by complete hemogram analysis | 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- School of Physical Education and Sports, University of Sao Paulo, São Paulo, São Paulo, Brazil